CLINICAL TRIAL: NCT00805246
Title: Identifying CT Imaging Biomarkers Associated With Prognosis of Pulmonary Embolism
Brief Title: Assessing the Prognosis of Pulmonary Embolism Using Clinical and Imaging Biomarkers (Retrospective & Prospective )
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kyongtae Ty Bae, M.D., Ph.D., Professor of Radiology and Bioengineering, University of Pittsburgh
Other Study IDs: HL095115; HL095115
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; PE; CT; Biomarker; Prognosis; Risk Prediction
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pulmonary Embolism (PE): Subjects diagnosed with PE by CT will be recruited.

SUMMARY:
Venous thromboembolism (VTE), which clinically manifests as deep vein thrombosis (DVT) and pulmonary embolism (PE), is a common but elusive illness that can cause significant disability and death if not promptly diagnosed and effectively treated. The annual incidence of VTE in the United States is estimated at 1 per 1000. Death occurs in approximately 12% of PE cases within 1 month of diagnosis. At present, clinical management of VTE and PE is hampered by gaps in our understanding of pathogenic mechanisms, the wide variety in patient populations, and incomplete understanding of the long term risks of recurrence and death. Given the complex presentation and risk associated with these conditions, proper risk assessment and subsequent prophylaxis for all at-risk patients is crucial. While clinical prediction rules have been recently developed to associate short-term risks and to stratify patients with acute PE, there is a dearth of objective biomarkers that can be related to the long-term prognosis of the disease. In addition to clinical information, clot burden is known to be strongly associated with clinical outcome of recurrent VTE. The quantification of clot burden requires imaging.

CT Pulmonary Angiography (CTPA) has been established as a reference imaging standard in the diagnosis of PE. In addition to its role as a superb diagnostic tool, CTPA contains a wealth of information including characteristics of the clot that may be used as biomarkers associated with prognosis of PE. The work proposed in this application takes advantage of widely available CTPA imaging biomarker data and extends and advances clinical PE risk prediction model to include long term (2-year) survival as well as the clinically important outcome of recurrence. The primary objective of this proposal is to develop and identify CTPA imaging biomarkers that are associated with short-term and long-term prognoses of patients who were positively diagnosed for PE by CT. The rationale for this proposal is that CT imaging is a rich source of imaging biomarkers that may be associated with prognosis of PE. This information will help advance our understanding of the risk and recurrence of PE and provide a new insight to prognosis and clinical management and treatment of PE. This proposed research is innovative in that we have developed new CT imaging biomarkers and designed a clinical trial to assess and validate the prognostic values of these biomarkers. Our central hypothesis is that CT imaging biomarkers are associated with the risk of death and recurrence in patients with PE. The specific aims of this proposal are: (1) to quantify and characterize pulmonary emboli (volume and distribution) and comorbid cardiovasculopulmonary findings from CT images of patients who were positively diagnosed for PE by CT; (2) to identify CT imaging biomarkers that are associated with the prognosis of patients who were positively diagnosed for PE by CT, and to develop risk prediction tools for death and recurrence; and (3) to prospectively validate the risk prediction tool, and identify whether the change in CT imaging biomarkers of PE after initiation of therapy improve the predictive ability for recurrence and death.

ELIGIBILITY:
Inclusion Criteria:

1. Adult > 18 years of age who either present to either hospital with acute PE or develop acute PE while admitted to the hospital diagnosed by CT
2. Capable of informed consent

Exclusion Criteria:

1. Contraindication to CT scanning
2. Cannot provide written informed consent.
3. Patients do not speak English, or have dementia and do not have a proxy who could participate in follow-up interviews.
4. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults > 18 years of age who either present to University of Pittsburgh Medical Center (UPMC) or Washington University in St. Louis hospitals with acute PE or develop acute PE while admitted to the hospital diagnosed by CT.
Sampling Method: Non-Probability Sample
Enrollment: 910 (Actual)
Dates: Start 2008-12; Primary Completion 2013-07 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The clinical and Imaging Biomarkers associated with Pulmonary Embolism (PE). | 5 years

SECONDARY OUTCOMES:
Pulmonary Embolism (PE) risk prediction rule. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca P. Link, Ph.D., Study Director — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania